CLINICAL TRIAL: NCT06946186
Title: Achieving Digital Equity for Health Improvement in a Virtual Senior Center
Brief Title: Virtual Senior Center
Acronym: VSC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Matthew Kreuter, Kahn Family Professor, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202408007; OT2HL158287 (NIH)
Record Dates: First submitted 2025-04-13; First posted 2025-04-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Social Isolation in Older Adults; Quality of Life (QOL); Activities of Daily Living
Keywords: digital access for older adults

STUDY DESIGN:
Intervention Model Description: Participants in 2 of the groups will be randomly assigned to receive the intervention immediately or in 6 month. The 3rd groups is naturally occurring comparison.
Masking Description: Though participants and investigators won't know condition of the randomized groups upon enrollment, they will know when they receive the GrandPad. The 3rd group will not be masked at any point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GrandPad1 (Experimental): This group will receive a GrandPad right away after they complete the baseline survey
  Interventions: Behavioral: Virtual Senior Center - GrandPad
- GrandPad2 - 6mo (Other): Delayed interventional. This group will receive a GrandPad after 6 months.
  Interventions: Behavioral: Virtual Senior Center - GrandPad
- Congregate (Active Comparator): This group will not receive a GrandPad but will get access to the Virtual Senior Center
  Interventions: Behavioral: Virtual Senior Center - No GrandPad

INTERVENTIONS:
Behavioral: Virtual Senior Center - GrandPad — The Virtual Senior Center engages older adults in programs and services online with the help of a GrandPad.
  Arms: GrandPad1; GrandPad2 - 6mo
Behavioral: Virtual Senior Center - No GrandPad — Participants will be given information to access the website when they are able from their own phone, tablet, or computer.
  Arms: Congregate

SUMMARY:
In a 3-group trial with randomization and follow-up for 12 months, we will compare use of the VSC as well as health and quality of life outcomes among 650 older adults in St. Louis who receive either: (1) home delivered meals AND a GrandPad; (2) home-delivered meals but no GrandPad for 6 months; and (3) in person meals at senior center but no GrandPad.

DETAILED DESCRIPTION:
The aims of the study are:

1. Recruit 650 older adults in St. Louis into the study - 400 home-delivered meal recipients and 250 receiving in-person meals at senior centers. Describe baseline differences between the two groups in use of senior center programming, technology access and use, and health and quality of life outcomes.
2. Randomly assign the 400 home-delivered meal recipients to get a GrandPad immediately (GP) or 6 months later (GP-6). Compare the GP and GP-6 groups to in-person meal recipients (IP) on: (A) VSC engagement at 6- and 12-month follow-up; and (B) health and quality of life outcomes at 6- and 12-month follow-up.
3. Examine longitudinal changes and hypothesized mediating pathways using 5 waves of data from baseline, 3-,6-,9- and 12-month follow-up. Specifically: (A) in the GP-6 group only, compare VSC engagement, health and quality of life outcomes at 6-month follow-up (a period in which they did not have a GrandPad) to 12-month follow-up (a period in which they did have a GrandPad); (B) examine 12-month trends in GrandPad and VSC engagement, health and quality of life outcomes within and across groups; and (C) test mediation of hypothesized explanatory variables from the study's conceptual framework to examine potential causal pathways for health and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current Home-delivered meal client with Aging Ahead

Exclusion Criteria:

* Under age 65

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The Social Isolation Scale in Older Adults (Nicholson et al., 2020; The Gerontologist) | 12 month
  This 6-item questionnaire measures the extent to which an individual feels socially unconnected, using 2 related constructs (3 items per construct): quantity of social contacts and sense of relationship. The response options for social contacts ranges from 1 (none) to 5 (6 or more) and the sense of relationship ranges from 1(strongly disagree) to 5 (strongly agree). The possible summed scores range from 6 to 30, with higher scores indicating less social isolation.

SECONDARY OUTCOMES:
Digital Social Participation (Anderberg et al., 2021; JMIR) | 12 month
  This 6-item questionnaire measures extent to which someone feels that digital technology is beneficial in their life. Response options range from 1 (strongly disagree) to 5 (strongly agree), so total summed scores range from 6 -30. A higher scores indicates more positive perceptions of digital technology.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kreuter, PhD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The raw survey response data including dates collected, as well as participant ID codes generated for this study will be shared in order to link the five waves of survey data as well as documentation of participation. All respondent identifiers (e.g., names, addresses) will be removed before sharing. Final de-identified intervention data and Common Survey 4 data will be shared with the CEAL (community engagement Alliance) Technical Assistance Team. Other CEAL researchers will be allowed to request common survey data.
  We will share all publicly accessible files on WashU Research Data, an institutional repository managed by the Washington University in St. Louis Libraries that uses a cloud-based hosted repository service called TIND as its platform. TIND is based on the open-source Invenio software developed at the research institute CERN to manage its own scholarly output. TIND uses an OAIS-compliant approach to preservation, with redundancy backup, conversion to archival file format
Supporting Information: Analytic Code
Time Frame: 3/31/28 - indefinitely
Access Criteria: Users must register with the repository and agree to the License specified for the project. This license will allow users to adapt and build upon the materials in any format for noncommercial purposes only and so long as attribution is given to the original creators and grant funding. Any adapted or new data formats and accompanying descriptions will also need to be publicly available under identical terms as the original. Additionally, the license will protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibit attempts to identify study participants, and require immediate reporting of any identification of study participant's identity. Data users also agree not to share or redistribute any data downloads.